CLINICAL TRIAL: NCT07171983
Title: A 2-Part, Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986454 in Participants With Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Safety, Tolerability, and Drug Levels of BMS-986454 in Participants With Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM055-1014
Record Dates: First submitted 2025-09-11; First posted 2025-09-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis (RA); Autoimmune Disease; Chronic Inflammatory Disease; Methotrexate-Inadequate Responders (MTX-IR)
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: Administration of BMS-986454 (Experimental)
  Interventions: Drug: BMS-986454
- Part A: Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Part B: Administration of BMS-986454 (Experimental)
  Interventions: Drug: BMS-986454
- Part B: Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986454 — Specified dose on specified days
  Arms: Part A: Administration of BMS-986454; Part B: Administration of BMS-986454
Other: Placebo — Specified dose on specified days
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and drug levels of BMS-986454 in participants with Rheumatoid Arthritis

ELIGIBILITY:
Inclusion Criteria:

* Participants with Rheumatoid Arthritis must have onset after age 18.
* Participants who meet 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria for RA.
* Participants must have evidence of swelling in at least 1 joint of the hand or wrist by clinical examination at screening and Day -1.
* Participants must have been an incomplete responder to prior methotrexate (MTX) treatment.

Exclusion Criteria:

* Participants must not have any significant medical condition, with the exception of Rheumatoid Arthritis (including but not limited to, neurological, GI, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders) that, in the Investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study.
* Participants must not have any condition aside from RA that confounds the ability to interpret data from the study.
* Participants must not have severe Rheumatoid Arthritis as assessed by Disease Activity Score 28 c-reactive protein (DAS28-CRP) at screening or Day -1.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-06-28 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 6 months
Number of participants with serious adverse events (SAEs) | Up to 6 months
Number of participants with physical examination findings | Up to 6 months
Number of participants with vital sign measurement findings | Up to 6 months
Number of participants with 12-lead electrocardiogram (ECG) findings | Up to 6 months
Number of participants with clinical laboratory test findings | Up to 6 months

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 6 months
Concentration at the end of a dosing interval (Ctau) | Up to 6 months
Trough observed plasma concentration (Ctrough) | Up to 6 months
Time of maximum observed concentration (Tmax) | Up to 6 months
Area under the curve over the dosing interval (AUC(TAU)) | Up to 6 months
Area under the serum concentration time curve extrapolated to infinite time (AUC(INF)) | Up to 6 months
Area under the serum concentration time curve from time zero to the last quantifiable concentration (AUC(0-T)) | Up to 6 months
Terminal-phase half-life (T-HALF) | Up to 6 months
Accumulation index of the area under the curve over the dosing interval (AI_AUC(TAU)) | Up to 6 months
Accumulation index of the maximum observed concentration (AI_Cmax) | Up to 6 months
Apparent total body clearance (CLT/F) | Up to 6 months
Apparent volume of distribution of terminal phase (Vz/F) | Up to 6 months
Number of participants with anti-drug antibody (ADA) formation | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- India (9):
  - Local Institution - 0006, Hyderabad, Andhra Pradesh
  - Local Institution - 0004, Ahmedabad, Gujarat
  - Local Institution - 0003, Bangalore, Karnataka
  - Local Institution - 0009, Mysuru, Karnataka
  - Local Institution - 0008, Nagpur, Maharashtra
  - Local Institution - 0005, Pune, Maharashtra
  - Local Institution - 0007, Bhubaneswar, Odisha
  - Local Institution - 0002, Hyderabad, Telangana
  - Local Institution - 0001, Secunderabad, Telangana

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html